CLINICAL TRIAL: NCT02717195
Title: Interventional, Randomised, Double-blind, Active-controlled, Fixed-dose Study of Lu AF35700 in Patients With Treatment-resistant Schizophrenia
Brief Title: Effect of Lu AF35700 in Patients With Treatment-resistant Schizophrenia
Acronym: DayBreak
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16159A; 2014-003569-12 (EudraCT Number)
Record Dates: First submitted 2016-03-11; First posted 2016-03-23 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Olanzapine; Lu AF35700

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prospective Confirmation (PC) Period (Experimental): Single (patient)-blinded treatment period with risperidone or olanzapine for 6 weeks
  Interventions: Drug: Risperidone; Drug: Olanzapine
- Double-blind Treatment (DBT) Period, Lu AF35700 10 mg (Experimental): Eligible patients from PC Period (based on criteria to which investigator and patient are blinded), will be randomly assigned (1:1:1) double-blind treatment in DBT Period, 10 weeks
  Interventions: Drug: Lu AF35700
- DBT Period, Lu AF35700 20 mg (Experimental): Eligible patients from PC Period (based on criteria to which investigator and patient are blinded), will be randomly assigned (1:1:1) double-blind treatment in DBT Period, 10 weeks
  Interventions: Drug: Lu AF35700
- DBT Period, Continued treatment from PC Period (Experimental): Eligible patients from PC Period (based on criteria to which investigator and patient are blinded), will be randomly assigned (1:1:1) double-blind treatment in DBT Period,10 weeks. Patients in this arm will continue with same the treatment and dose as at last visit of PC Period
  Interventions: Drug: Risperidone; Drug: Olanzapine

INTERVENTIONS:
Drug: Risperidone — 4-6 mg/day, encapsulated tablets, orally
  Arms: DBT Period, Continued treatment from PC Period; Prospective Confirmation (PC) Period
Drug: Olanzapine — 15-20 mg/day, encapsulated tablets, orally
  Arms: DBT Period, Continued treatment from PC Period; Prospective Confirmation (PC) Period
Drug: Lu AF35700 — 10 mg/day, encapsulated tablets, orally
  Arms: Double-blind Treatment (DBT) Period, Lu AF35700 10 mg
Drug: Lu AF35700 — 20 mg/day, encapsulated tablets, orally
  Arms: DBT Period, Lu AF35700 20 mg

SUMMARY:
To evaluate the efficacy of 10 and 20 mg/day of Lu AF35700 on schizophrenia symptoms in patients with treatment-resistant schizophrenia (TRS)

DETAILED DESCRIPTION:
The study consists of a Screening Period (3 weeks), a single-blind Prospective Confirmation (PC) Period (6 weeks), a Double-blind Treatment (DBT) Period (10 weeks), and a Safety Follow-up Period (6 weeks).

Patients who did not fulfil the randomization criteria for the DBT Period, were withdrawn from the study after the PC period.

Patients who fulfilled the randomization criteria for the DBT Period, continued into the DBT Period and were randomized into one of 3 treatment arms (1:1:1) with either Lu AF35700 10 mg/day, Lu AF35700 20 mg/day or to continue the treatment allocated in PC Period (olanzapine or risperidone) at the dose set at last visit of PC Period. This mean that approximately one third of the confirmed treatment-resistant patients were randomised back to the failed treatment used in the PC Period.

Data was not collected separately for the DBT Olanzapine and DBT Risperidone participants, and there was no intent to compare Lu AF35700 to each drug separately.

ELIGIBILITY:
Inclusion Criteria:

* The patient has schizophrenia, diagnosed according to DSM-5(TM) (Diagnostic and Statistical Manual of Mental Disorders) and confirmed by the Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorders
* The patient is either an inpatient at a psychiatric setting or outpatient consulting a psychiatrist.
* Patients should be treated with adequate dose(s) and agent(s) of antipsychotic treatment for at least 2 weeks prior to Screening
* The patient has failed to show an adequate response in the level of psychotic symptoms despite at least one documented treatment trial with an adequate dose of an antipsychotic agent prescribed for an adequate time (at least lasting for 6 weeks) during 2 years prior to Screening. The failure to respond to the current antipsychotic treatment trial may be considered a retrospective failed treatment, if the patient was treated for 6 weeks with adequate dose(s) and agent(s)
* The patient has a PANSS total score of ≥80 and a score of ≥4 on at least 2 of the following PANSS items (at Screening and at the first visit of Period A)
* The patient has a CGI-S score of ≥4 at Screening and at the first visit of Period A

Exclusion Criteria:

* The patient has any current primary psychiatric disorder other than schizophrenia as assessed by the Mini International Neuropsychiatric Interview (MINI)
* The patient is experiencing an acute exacerbation of his/her psychotic symptoms
* The patient has not responded to treatment with clozapine

Other protocol defined inclusion and exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1098 (Actual)
Dates: Start 2016-04; Primary Completion 2018-08-30 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (147):
- United States (49):
  - US1018, Bellflower, California
  - US1041, Cerritos, California
  - US1062, Costa Mesa, California
  - US1463, Culver City, California
  - US1104, Garden Grove, California
  - US1118, Glendale, California
  - US1114, National City, California
  - US1452, Oceanside, California
  - US1459, Oceanside, California
  - US1399, Orange, California
  - US1368, Orange, California
  - US1391, San Bernardino, California
  - US1464, Santa Ana, California
  - US1384, Sherman Oaks, California
  - US1392, Torrance, California
  - US1396, Washington D.C., District of Columbia
  - US1395, Bradenton, Florida
  - US1253, Jacksonville, Florida
  - US1130, Miami, Florida
  - US1318, North Miami, Florida
  - US1129, North Miami, Florida
  - US1402, Oakland Park, Florida
  - US1229, Orange City, Florida
  - US1453, Tampa, Florida
  - US1403, Atlanta, Georgia
  - US1009, Atlanta, Georgia
  - US1442, Decatur, Georgia
  - US1046, Chicago, Illinois
  - US1423, Hoffman Estates, Illinois
  - US1398, Shreveport, Louisiana
  - US1404, Shreveport, Louisiana
  - US1086, Flowood, Mississippi
  - US1444, Las Vegas, Nevada
  - US1426, Berlin, New Jersey
  - US1454, Marlton, New Jersey
  - US1405, Glen Oaks, New York
  - US1244, Jamaica, New York
  - US1394, New York, New York
  - US1416, New York, New York
  - US1171, Rochester, New York
  - US1190, Staten Island, New York
  - US1390, Charlotte, North Carolina
  - US1401, Charlotte, North Carolina
  - US1441, Hickory, North Carolina
  - US1124, Norristown, Pennsylvania
  - US1319, Charleston, South Carolina
  - US1451, Austin, Texas
  - US1065, Dallas, Texas
  - US1443, Fort Worth, Texas
- Bulgaria (12):
  - BG1030, Burgas
  - BG1028, Kazanlak
  - BG1003, Lovech
  - BG1032, Pazardzhik
  - BG1008, Plovdiv
  - BG1024, Sofia
  - BG1026, Sofia
  - BG1022, Tserova Koria
  - BG1033, Varna
  - BG1034, Varna
  - BG1029, Veliko Tarnovo
  - BG1027, Vratsa
- Canada (6):
  - CA1017, Chatham
  - CA1034, Kingston
  - CA1003, Montreal
  - CA1033, Montreal
  - CA1029, Penticton
  - CA1039, Québec
- Czechia (5):
  - CZ1023, Brno
  - CZ1032, Brno
  - CZ1037, Hostivice
  - CZ1013, Lnáře
  - CZ1038, Prague
- Estonia (3):
  - EE1016, Pärnu
  - EE1007, Tallinn
  - EE1017, Viljandi
- Finland (3):
  - FI1032, Espoo
  - FI1030, Kuopio
  - FI1027, Turku
- Mexico (10):
  - MX1024, Durango
  - MX1011, Guadalajara
  - MX1021, Guadalajara
  - MX1022, Guadalajara
  - MX1020, México
  - MX1005, Monterrey
  - MX1007, Monterrey
  - MX1015, Monterrey
  - MX1016, Monterrey
  - MX1018, San Luis Potosí City
- Poland (9):
  - PL1025, Bełchatów
  - PL1043, Bialystok
  - PL1026, Gorlice
  - PL1060, Lodz
  - PL1027, Lublin
  - PL1058, Pruszcz Gdański
  - PL1061, Pruszków
  - PL1059, Torun
  - PL1051, Wroclaw
- Romania (4):
  - RO1024, Bucharest
  - RO1022, Campulung Muscel
  - RO1025, Sibiu
  - RO1004, Târgu Mureş
- Russia (14):
  - RU1021, Nikol’skoye, Gatchinckiy District
  - RU1009, Arkhangelsk
  - RU1006, Moscow
  - RU1051, Moscow
  - RU1055, Moscow
  - RU1023, Saint Petersburg
  - RU1028, Saint Petersburg
  - RU1030, Saint Petersburg
  - RU1031, Saint Petersburg
  - RU1049, Saint Petersburg
  - RU1052, Saint Petersburg
  - RU1053, Saint Petersburg
  - RU1056, Saint Petersburg
  - RU1050, Yaroslavl
- Serbia (8):
  - RS1008, Belgrade
  - RS1010, Belgrade
  - RS1012, Belgrade
  - RS1011, Kragujevac
  - RS1016, Kragujevac
  - RS1017, Kragujevac
  - RS1003, Niš
  - RS1009, Novi Kneževac
- Slovakia (5):
  - SK1014, Bratislava
  - SK1024, Bratislava
  - SK1015, Rožňava
  - SK1025, Svidník
  - SK1026, Zlaté Moravce
- Spain (5):
  - ES1047, Barcelona
  - ES1012, Madrid
  - ES1008, Málaga
  - ES1048, Oviedo
  - ES1049, Zamora
- Ukraine (14):
  - UA1019, Dnipropetrovsk
  - UA1017, Kharkiv
  - UA1022, Kharkiv
  - UA1031, Kharkiv
  - UA1035, Kharkiv
  - UA1028, Kherson
  - UA1029, Kherson
  - UA1027, Kiev
  - UA1030, Kiev
  - UA1033, Lviv
  - UA1020, Odesa
  - UA1032, Odesa
  - UA1001, Poltava
  - UA1036, Vinnitsa

REFERENCES:
- [Derived] Kane JM, Kinon BJ, Forray C, Such P, Mittoux A, Lemming OM, Hertel P, Howes OD; DayBreak and Debut study investigators. Efficacy and safety of Lu AF35700 in treatment-resistant schizophrenia: A randomized, active-controlled trial with open-label extension. Schizophr Res. 2022 Oct;248:271-278. doi: 10.1016/j.schres.2022.09.012. Epub 2022 Sep 14. PMID 36115192

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who did not fulfil the randomization criteria for the DBT Period, were withdrawn from the study after the PC period. Patients who fulfilled the randomization criteria for the DBT Period, continued into the DBT Period. Patients randomized into the DBT period with risperidone or olanzapine were analyzed as one arm independent of treatment.
Groups:
- Prospective Confirmation (PC) Period, Risperidone: Single (patient)-blinded treatment period with risperidone or olanzapine for 6 weeks
  Risperidone: 4-6 mg/day, encapsulated tablets, orally
- PC Period, Olanzapine: Single (patient)-blinded treatment period with risperidone or olanzapine for 6 weeks
  Olanzapine: 15-20 mg/day, encapsulated tablets, orally
- Double-blind Treatment (DBT) Period, Lu AF35700 10 mg: Lu AF35700: 10 mg/day, encapsulated tablets, orally for 10 weeks
- DBT Period, Lu AF35700 20 mg: Lu AF35700: 20 mg/day, encapsulated tablets, orally for 10 weeks
- DBT Period, Continued Treatment From PC Period: Patients in this arm will continue the treatment allocated in the PC Period at the dose set at last visit of the PC Period. The analysis is made independent on which treatment the patient was on (risperidone or olanzapine)
Period: Prospective Confirmation (PC) Period
Arm/Group | Prospective Confirmation (PC) Period, Risperidone | PC Period, Olanzapine | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Started | 711 | 387 | 0 | 0 | 0
Completed | 421 | 276 | 0 | 0 | 0
Not Completed | 290 | 111 | 0 | 0 | 0
Not completed — Adverse Event | 19 | 7 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0 | 0
Not completed — Non-compliance with IMP | 7 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 43 | 12 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 4 | 0 | 0 | 0
Not completed — Did not fulfill rand criteria for DBT | 189 | 75 | 0 | 0 | 0
Not completed — Enrolled but not treated | 3 | 3 | 0 | 0 | 0
Not completed — Lack of results for blood levels | 1 | 0 | 0 | 0 | 0
Not completed — Technical error | 1 | 0 | 0 | 0 | 0
Not completed — Patient decision | 5 | 2 | 0 | 0 | 0
Not completed — Low level of drug in the blood | 1 | 0 | 0 | 0 | 0
Not completed — Change of place of residence | 1 | 0 | 0 | 0 | 0
Not completed — Apato Abulcasis Syndrome | 0 | 1 | 0 | 0 | 0
Not completed — Investigator decision | 2 | 1 | 0 | 0 | 0
Not completed — Subject took exclusionary medication | 0 | 1 | 0 | 0 | 0
Not completed — Sub therapeutic blood levels Olanzapine | 1 | 0 | 0 | 0 | 0
Not completed — Positive Urine Drug Screen | 0 | 1 | 0 | 0 | 0
Not completed — Duplicate subject | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor requested | 0 | 1 | 0 | 0 | 0
Not completed — Patient fraud with payment | 1 | 0 | 0 | 0 | 0
Not completed — Noncompliance with protocol | 1 | 0 | 0 | 0 | 0
Period: Double-blind Treatment (DBT) Period
Arm/Group | Prospective Confirmation (PC) Period, Risperidone | PC Period, Olanzapine | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Started | 0 | 0 | 235 | 232 | 230
Completed | 0 | 0 | 198 | 188 | 200
Not Completed | 0 | 0 | 37 | 44 | 30
Not completed — Adverse Event | 0 | 0 | 10 | 11 | 8
Not completed — Lack of Efficacy | 0 | 0 | 6 | 9 | 2
Not completed — Non-compliance with IMP | 0 | 0 | 4 | 3 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 14 | 13 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 2
Not completed — Enrolled but not treated | 0 | 0 | 1 | 0 | 0
Not completed — Patient decision | 0 | 0 | 0 | 2 | 2
Not completed — Investigator decision | 0 | 0 | 0 | 1 | 1
Not completed — Family circumstances | 0 | 0 | 0 | 0 | 1
Not completed — Change of residence | 0 | 0 | 0 | 1 | 1
Not completed — Needed antidepressant medication | 0 | 0 | 0 | 0 | 1
Not completed — Psychosocial issues | 0 | 0 | 1 | 0 | 0
Not completed — Patient missed required visits | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-randomized Patients: Patients not randomized into the double-blind treatment period, i.e. withdrawn from the study during or after the PC period, were analyzed as one arm independent of treatment.
- DBT Period, Continued Treatment From PC Period: Patients in this arm continued with the same treatment and dose as at the last visit of the PC Period. Patients randomized into the DBT period with risperidone or olanzapine were analyzed as one arm independent of treatment.
- Total: Total of all reporting groups
Arm/Group | Non-randomized Patients | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period | Total
Number analyzed (Participants) | 401 | 235 | 232 | 230 | 1098
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11.05) | 42.6 (12.14) | 42.3 (11.44) | 43.2 (11.19) | 43 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 91 | 94 | 89 | 421
  Male | 254 | 144 | 138 | 141 | 677
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 6 | 10 | 8 | 59
  Not Hispanic or Latino | 224 | 46 | 42 | 45 | 357
  Unknown or Not Reported | 142 | 183 | 180 | 177 | 682
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 4 | 1 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 172 | 36 | 33 | 34 | 275
  White | 186 | 176 | 179 | 178 | 719
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 36 | 22 | 19 | 17 | 94
PANSS total score [Mean (Standard Deviation); unit: units on a scale] — PANSS total score administered by the investigator. It included 3 sub-scales with a total of 30 items that evaluated the Positive Symptoms subscale, the Negative Symptoms subscale, the General Psychopathology subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). PANSS total score was calculated as sum of all the items on the scale and ranged from 30 to 210. A higher score corresponded to a worse severity of schizophrenia.
  units on a scale | 97.25 (11.21) | 96.96 (9.17) | 98.23 (9.29) | 98.40 (9.84) | 97.6 (10.12)
CGI-S score [Mean (Standard Deviation); unit: units on a scale] — CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients). Higher scores indicate worsening.
  units on a scale | 4.82 (0.60) | 4.88 (0.59) | 5.00 (0.57) | 4.90 (0.53) | 4.89 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization to Week 10 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: PANSS total score administered by the investigator. It included 3 sub-scales with a total of 30 items that evaluated the Positive Symptoms subscale, the Negative Symptoms subscale, the General Psychopathology subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). PANSS total score was calculated as sum of all the items on the scale and ranged from 30 to 210. A higher score corresponded to a worse severity of schizophrenia.
Time Frame: From Randomization to Week 10
Population: Only patients randomized to receive double-blind treatment in the DBT Period are analysed. Patients randomized into the DBT period with risperidone or olanzapine were analyzed as one arm independent of treatment. Overall Number of Participants Analysed is number of patients in the FAS with a week 10 observation.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- DBT Period, Continued Treatment From PC Period: Patients in this arm will continue with the same treatment and dose as at the last visit of the PC Period (olanzapine or risperidone)
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 201 | 189 | 202
units on a scale | -10.01 (0.96) | -8.22 (0.98) | -9.90 (0.97)
Statistical Analysis 1: Comparison: Double-blind Treatment (DBT) Period, Lu AF35700 10 mg vs DBT Period, Continued Treatment From PC Period; The mean changes from Randomization in PANSS total score was analysed using a MMRM approach. The model included the fixed, categorical effects of treatment, country, week, treatment-by-week interaction, PC Period treatment, PC Period treatment-by-week interaction, and the continuous covariates of Randomization score and Randomization score-by-week interaction with an unstructured covariance structure to model the within-patient errors; Test type: Superiority; p = 0.9196, Mixed model repeated measures — Multiplicity adjustment was planned for the testing of the primary enpoint, but was not applied since all p-values>0.05; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-2.37 to 2.13]
Statistical Analysis 2: Comparison: DBT Period, Lu AF35700 20 mg vs DBT Period, Continued Treatment From PC Period; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1474, Mixed model repeated measures — Multiplicity adjustment was planned for the testing of the primary endpoint, but was not applied since all p-values>0.05; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [-0.59 to 3.94]

2. Secondary Outcome: Change From Randomization to Week 10 in PSP Total Personal and Social Performance (PSP) Total Score
Description: PSP is a clinician-rated scale designed and validated to measure a patient's current level of social functioning. It consists of 4 items: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviours. Each items were assessed on a 6-point scale, from 1 (absent) to 6 (very severe). PSP score was calculated as sum of all the items on the scale and ranged from 4 to 100. A higher score represents more severe functional impairment.
Time Frame: From Randomization to Week 10
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 204 | 197 | 203
units on a scale | 4.90 (0.96) | 3.23 (0.98) | 3.94 (0.98)
Statistical Analysis 1: Comparison: Double-blind Treatment (DBT) Period, Lu AF35700 10 mg vs DBT Period, Continued Treatment From PC Period; The mean changes from Randomization in PSP score was analysed using a MMRM approach. The model included the fixed, categorical effects of treatment, country, week, treatment-by-week interaction, PC Period treatment, PC Period treatment-by-week interaction, and the continuous covariates of Randomization score and Randomization score-by-week interaction with an unstructured covariance structure to model the within-patient errors; Test type: Superiority; p = 0.2998, Mixed model repeated measures — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-0.86 to 2.78]
Statistical Analysis 2: Comparison: DBT Period, Lu AF35700 20 mg vs DBT Period, Continued Treatment From PC Period; The mean changes in PSP score was analysed using a MMRM approach. The model included the fixed, categorical effects of treatment, country, week, treatment-by-week interaction, PC Period treatment, PC Period treatment-by-week interaction, and the continuous covariates of Randomization score and Randomization score-by-week interaction with an unstructured covariance structure to model the within-patient errors; Test type: Superiority; p = 0.4478, Mixed model repeated measures — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-2.54 to 1.12]

3. Secondary Outcome: Change From Randomization to Week 10 in Global Clinical Impression - Severity of Illness (CGI-S) Score
Description: CGI-S provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients). Higher scores indicate worsening.
Time Frame: From Randomization to Week 10
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 232 | 231 | 228
units on a scale | -0.59 (0.06) | -0.54 (0.06) | -0.57 (0.06)

4. Secondary Outcome: Response at Week 10, Defined as ≥20% Reduction in PANSS Total Score, PANSS (Positive and Negative Syndrome Scale) Total Score ≤70, CGI-S (Clinical Global Impression Scale - Severity of Illness) Score <4
Description: PANSS total score administered by the investigator. It included 3 sub-scales with a total of 30 items that evaluated the Positive Symptoms subscale, the Negative Symptoms subscale, the General Psychopathology subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). PANSS total score was calculated as sum of all the items on the scale and ranged from 30 to 210. A higher score corresponded to a worse severity of schizophrenia. A reduction in score indicates improvement.
  The Clinical Global Impression scale - severity of illness (CGI-S) is administered by the investigator. The patient is rated on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients). A reduction in scale indicates improvement.
Time Frame: From Randomization to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 201 | 189 | 202
Participants | 21 | 18 | 12

5. Secondary Outcome: Response at Week 10, Defined as ≥20% Reduction in Positive and Negative Syndrome Scale (PANSS) Total Score From Randomization
Description: PANSS total score administered by the investigator. It included 3 sub-scales with a total of 30 items that evaluated the Positive Symptoms subscale, the Negative Symptoms subscale, the General Psychopathology subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). PANSS total score was calculated as sum of all the items on the scale and ranged from 30 to 210. A higher score corresponded to a worse severity of schizophrenia. A reduction in score indicates improvement.
Time Frame: From Randomization to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 201 | 189 | 202
Participants | 82 | 59 | 77

6. Secondary Outcome: Response at Week 10, Defined as ≥30% Reduction in PANSS Total Score From Randomization
Description: Positive and Negative Syndrome Scale (PANSS) total score administered by the investigator. It included 3 sub-scales with a total of 30 items that evaluated the Positive Symptoms subscale, the Negative Symptoms subscale, the General Psychopathology subscale. Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). PANSS total score was calculated as sum of all the items on the scale and ranged from 30 to 210. A higher score corresponded to a worse severity of schizophrenia. A reduction in score indicates improvement.
Time Frame: From Randomization to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 201 | 189 | 202
Participants | 42 | 30 | 45

7. Secondary Outcome: Response at Week 10, Defined as ≥40% Reduction in Positive and Negative Syndrome Scale (PANSS) Total Score From Randomization
Description: as for outcome 5
Time Frame: From Randomization to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 201 | 189 | 202
Participants | 23 | 15 | 16

8. Secondary Outcome: Response at Week 10, Defined as ≥50% Reduction in Positive and Negative Syndrome Scale (PANSS) Total Score From Randomization
Description: as for outcome 5
Time Frame: From Randomization to Week 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
Number analyzed (Participants) | 201 | 189 | 202
Participants | 10 | 4 | 6

ADVERSE EVENTS:
Time Frame: 22 weeks
Groups:
- Prospective Confirmation (PC) Period, Risperidone; PC Period, Olanzapine: Patients not randomized to double-blind treatment
- Double Blind Treatment (DBT) Period, Lu AF35700 10 mg: Lu AF35700: 10 mg/day, encapsulated tablets, orally for 10 weeks
- DBT Period, Continued Treatment From PC Period: Patients in this arm continued with the same treatment and dose as at the last visit of the PC Period. This arm is analyzed as one single treatment arm independent on which treatment was administered (olanzapine or risperidone).
Arm/Group | Prospective Confirmation (PC) Period, Risperidone | PC Period, Olanzapine | Double Blind Treatment (DBT) Period, Lu AF35700 10 mg | DBT Period, Lu AF35700 20 mg | DBT Period, Continued Treatment From PC Period
All-Cause Mortality (participants affected / at risk) | 0/708 | 0/384 | 0/234 | 0/232 | 1/230
Serious Adverse Events (participants affected / at risk) | 14/708 | 7/384 | 6/234 | 5/232 | 5/230
Other Adverse Events (participants affected / at risk) | 60/708 | 45/384 | 20/235 | 40/232 | 25/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Confirmation (PC) Period, Risperidone (N=708) | PC Period, Olanzapine (N=384) | Double Blind Treatment (DBT) Period, Lu AF35700 10 mg (N=234) | DBT Period, Lu AF35700 20 mg (N=232) | DBT Period, Continued Treatment From PC Period (N=230)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vascular stent thrombosis (General disorders) | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 5 | 1 | 1 | 2 | 2
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 2 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Social stay hospitalisation (Social circumstances) | 1 | 1 | 0 | 0 | 0
Psychosocial support (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Confirmation (PC) Period, Risperidone (N=708) | PC Period, Olanzapine (N=384) | Double Blind Treatment (DBT) Period, Lu AF35700 10 mg (N=235) | DBT Period, Lu AF35700 20 mg (N=232) | DBT Period, Continued Treatment From PC Period (N=230)
Weight increased (Investigations) | 5 | 1 | 8 | 19 | 11
Headache (Nervous system disorders) | 24 | 16 | 11 | 15 | 10
Somnolence (Nervous system disorders) | 34 | 30 | 3 | 9 | 4
Akathisia (Nervous system disorders) | 36 | 8 | 3 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02717195/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT02717195/SAP_001.pdf